CLINICAL TRIAL: NCT03365518
Title: Innovations in the Treatment of Sexual Dysfunction and Couple Intimacy After Prostate Cancer: A Randomized Trial of Mindfulness Versus Cognitive Behavioural Therapy
Brief Title: Innovations in the Treatment of Sexual Health Post Prostate Cancer Treatment: Comparing Mindfulness vs. CBT
Acronym: INTROSPPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Prostate Centre (Other)
Responsible Party: Principal Investigator, Lori Brotto, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H17-02247; D2017-1893 (Other Grant/Funding Number: Movember Discovery Grant/Prostate Cancer Canada)
Record Dates: First submitted 2017-12-01; First posted 2017-12-07 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer; Sexual Dysfunctions, Psychological; Sexual Dysfunction, Physiological; Sexual Dysfunction Male; Relationships, Marital; Prostatic Neoplasms
Keywords: Psychological Treatment; Intimacy; Cognitive Behavioural Therapy; Cognitive Behavioral Therapy; Mindfulness; Group Therapy; Couples Therapy
MeSH Terms: conditions — Prostatic Neoplasms; Sexual Dysfunctions, Psychological; Sexual Dysfunction, Physiological | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Behavioural Therapy (CBT) (Experimental): Treatment will consist of a 4-week group lead by a trained clinician. Sessions are 2 hours in length and take place in consecutive weeks, with daily homework recommended between sessions.
  Interventions: Behavioral: Cognitive Behavioural Therapy (CBT)
- Mindfulness-Based Therapy (Experimental): Treatment will consist of a 4-week group lead by a trained clinician. Sessions are 2 hours in length and take place in consecutive weeks, with daily homework recommended between sessions.
  Interventions: Behavioral: Mindfulness-Based Therapy
- Control - Usual Care (No Intervention): Participants who are randomized to the control group will not receive mindfulness or CBT treatment. They will proceed with the course of treatment they were receiving prior to enrollment in the study. As resources for couples dealing with changes to their sexual lives after prostate cancer are limited, it is anticipated that the majority of these patients will have no treatment targeting sexual intimacy during the 6-week period between completing the first and second questionnaire.
  Those randomized to the "control" group will have the opportunity to be randomized to one of the treatment groups following their third and final questionnaire if they wish. In this case, they will be issued an additional participant ID within one of the treatment groups.

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy (CBT) — Sessions consist of CBT tools as well as sex therapy techniques and education. The CBT treatment was adapted from the mindfulness-based treatment, but all mentions of mindfulness have been replaced with CBT principles. The therapeutic content presented in this treatment arm is manualized.
  Arms: Cognitive Behavioural Therapy (CBT)
Behavioral: Mindfulness-Based Therapy — The mindfulness-based treatment was developed based on pre-existing mindfulness-based cognitive therapy treatment groups for sexual dysfunction developed by Dr. Lori Brotto at the University of British Columbia Sexual Health Laboratory, mindfulness in Sex therapy and Intimate Relationships (MSIR) treatment group developed by Kocsis and Newbury-Helps (2016), and expert input. Sessions consist of mindfulness-based training as well as sex therapy techniques and education. The therapeutic content presented in this treatment arm is manualized.
  Arms: Mindfulness-Based Therapy

SUMMARY:
Up to 90% of men experience sexual difficulties after receiving treatment for prostate cancer (PC), which can negatively affect their intimate relationships and overall quality of life. In this randomized clinical trial, the investigators will assess and compare two evidence-based treatments, mindfulness-based therapy and cognitive behavioral therapy (CBT), for couples with sexual complaints following PC treatment to controls who will receive no intervention.

DETAILED DESCRIPTION:
This randomized clinical trial is designed to assess and compare efficacy of two treatment manuals for couples with sexual difficulties secondary to PC treatment: mindfulness-based therapy and CBT. A third arm, where couples receive no intervention will act as a control group. Those randomized to the "control" group will have the opportunity to be randomized to one of the treatment groups following their third and final questionnaire if they wish.

Men and their partners will be invited to participate through the Vancouver Prostate Centre's Prostate Cancer Supportive Care Program (PCSC) at Vancouver General Hospital.

Eligible couples will be randomized to either: 4 consecutive weeks of mindfulness-based therapy, CBT, or no intervention (4-6 couples in each treatment group at a time). All participants will complete an online questionnaire package to assess primary, secondary, and tertiary outcomes at the time of study enrollment or baseline (Time 1). All participants will be invited to complete a Time 2 questionnaire once approximately 6 weeks after they complete the Time 1 questionnaire (for couples randomized to the treatment arms, this will be immediately post-treatment). Finally, all participants will be invited to complete the Time 3 follow up questionnaire 6 months after they complete the Time 2 (post-treatment) questionnaire.

Endpoints will assess effects on intimacy and overall Quality of Life. Additional endpoints of other factors affecting improvement (i.e., moderators like personality and treatment adherence) will be assessed. The investigators predict improvements in both mindfulness-based and cognitive behavioural therapy treatments; moderators will provide insights into which participants benefit most from each treatment arm.

Moreover, in order to improve understanding of the lived experience of patients who take part in the treatment groups or control arm, this study will invite all participants to take part in an exit interview after their Time 2 (post-treatment) questionnaire is completed. A research team member who was not a treatment facilitator will conduct the exit interviews. This information will then be transcribed and used for qualitative data analyses.

ELIGIBILITY:
Inclusion Criteria:

* Currently in a relationship that has lasted longer than 1 year
* Both members of the couple are at least 19 years of age or older
* (At least) one member of the couple has a history of prostate cancer diagnosis
* The same member of the couple underwent treatment (e.g., radical prostatectomy, radiation therapy, Androgen Deprivation Therapy) for their prostate cancer or is on active surveillance
* The member of the couple who underwent treatment for prostate cancer is experiencing distress related to his current level of intimacy/sexual well-being
* Both members of the couple are willing and able to comply with all study procedures and be available for the duration of the study. Commitment includes a total of 5.5 hours per week in sessions and daily homework over the 4-week period of the treatment program for those randomized to receive treatment
* Both members of the couple are fluent in English

Exclusion Criteria:

* Have a current health condition (e.g., severe cardiovascular health problems, unmanaged diabetes mellitus), physical disability and/or a significant, unmanaged major mental illness (e.g., unmanaged bipolar disorder, psychosis) that would interfere with self- or partnered-sexual activities, or the individual's ability to attend group sessions or complete home assignments

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Change in relationship satisfaction | Baseline and Post Treatment (6 weeks)
  Adapted dyadic adjustment scale (A-DAS). The A-DAS is a validated, 7-item measure that assesses relationship adjustment. Total scores range from 0-36 with higher scores indicating greater dyadic adjustment.
Change in relationship satisfaction | Baseline and Follow Up (6 months)
  Adapted dyadic adjustment scale (A-DAS). The A-DAS is a validated, 7-item measure that assesses relationship adjustment. Total scores range from 0-36 with higher scores indicating greater dyadic adjustment.
Change in sexual satisfaction/distress | Baseline and Post Treatment (6 weeks)
  Female sexual distress scale - revised (FSDS-R). The FSDS-R is a 13-item measure that assesses sexual distress. Although named for its use with women, this measure has been validated as a measure of sexual distress in women and men. Each item is rated on a scale of 0-4. The total score is a summation, ranging from 0 to 52, and provides a measure of sexual distress in which higher scores represent higher levels of sexual distress.
Change in sexual satisfaction/distress | Baseline and Follow Up (6 months)
  Female sexual distress scale - revised (FSDS-R). The FSDS-R is a 13-item measure that assesses sexual distress. Although named for its use with women, this measure has been validated as a measure of sexual distress in women and men. Each item is rated on a scale of 0-4. The total score is a summation, ranging from 0 to 52, and provides a measure of sexual distress in which higher scores represent higher levels of sexual distress.
Change in sexual functioning (one of three different questionnaires depending on the participant's demographics) | Baseline and Post Treatment (6 weeks)
  International Index of Erectile Functioning (IIEF) is a 15-item self-reported scale of men's sexual functioning. The scale has five domains: Erectile Function, Intercourse Satisfaction; Orgasmic Function, Overall Satisfaction, and Sexual Desire with ranges 1-30, 0-15, 0-10, 2-10, and 2-10 respectively. Total scores (sum) range from 5-75. Lower domain and total scores denote lower sexual function.
  OR International Index of Erectile Functioning for Men who have sex with men (IIEF-MSM) is a 22-item measure of sexual function. Total scores (sum) range from 0-95; lower scores indicate lower sexual function.
  OR Female Sexual Functioning Index (FSFI) is a 19-item measure of self-reported sexual dysfunction in women. The scale includes six domains with the following ranges: 1.2-6 for desire; 0-6 for arousal, lubrication, orgasm, and pain; and 0.8-6 satisfaction. Total scores (sum) range from 2 to 36. Lower domain and total scores indicate lower sexual functioning.
Change in sexual functioning (one of three different questionnaires depending on the participant's demographics) | Baseline and Follow Up (6 months)
  International Index of Erectile Functioning (IIEF) is a 15-item self-reported scale of men's sexual functioning. The scale has five domains: Erectile Function, Intercourse Satisfaction; Orgasmic Function, Overall Satisfaction, and Sexual Desire with ranges 1-30, 0-15, 0-10, 2-10, and 2-10 respectively. Total scores (sum) range from 5-75. Lower domain and total scores denote lower sexual function.
  OR International Index of Erectile Functioning for Men who have sex with men (IIEF-MSM) is a 22-item measure of sexual function. Total scores (sum) range from 0-95; lower scores indicate lower sexual function.
  OR Female Sexual Functioning Index (FSFI) is a 19-item measure of self-reported sexual dysfunction in women. The scale includes six domains with the following ranges: 1.2-6 for desire; 0-6 for arousal, lubrication, orgasm, and pain; and 0.8-6 satisfaction. Total scores (sum) range from 2 to 36. Lower domain and total scores indicate lower sexual functioning.
Change in sexual behaviours | Baseline and Post Treatment (6 weeks)
  Sexual activity scale. This is a questionnaire developed by the study lead that asks individuals to indicate whether they engaged in a range of sexual activities over 3 time-periods: (a) ever, (b) since their/their partner's prostate cancer surgery, and (c) in the past 4 weeks. There are 15 items on this scale which can be indicated over the three time periods mentioned previously. By tallying the categorical answers (yes or no), total scores can range from 0 to 45 with higher scores indicating greater sexual activity engaged. Subset scores at each time point range from 0-15 and indicate sexual activity in the same way as the total score.
Change in sexual behaviours | Baseline and Follow Up (6 months)
  Sexual activity scale. This is a questionnaire developed by the study lead that asks individuals to indicate whether they engaged in a range of sexual activities over 3 time-periods: (a) ever, (b) since their/their partner's prostate cancer surgery, and (c) in the past 4 weeks. There are 15 items on this scale which can be indicated over the three time periods mentioned previously. By tallying the categorical answers (yes or no), total scores can range from 0 to 45 with higher scores indicating greater sexual activity engaged. Subset scores at each time point range from 0-15 and indicate sexual activity in the same way as the total score.

SECONDARY OUTCOMES:
Change in psychological well-being | Baseline and Post Treatment (6 weeks)
  Hospital Anxiety and Depression Scale (HADS). The HADS is a validated, 14-item measure of depression and anxiety. Total scores range from 0-42, composed of the sum of two sub-scales for anxiety and depression both ranging from 0-21. Higher scores indicate higher levels of anxiety and/or depression symptoms.
Change in psychological well-being | Baseline and Follow Up (6 months)
  Hospital Anxiety and Depression Scale (HADS). The HADS is a validated, 14-item measure of depression and anxiety. Total scores range from 0-42, composed of the sum of two sub-scales for anxiety and depression both ranging from 0-21. Higher scores indicate higher levels of anxiety and/or depression symptoms.
Change in distress | Baseline and Post Treatment (6 weeks)
  Distress Thermometer. The distress thermometer is a single-item distress screening scale, which has been shown to be a valid measure of cancer-specific distress among prostate cancer patients and their partners. Participants indicate their current level of distress on an 11-point scale from 0-10 with 0 being no distress and 10 being extreme distress.
Change in distress | Baseline and Follow Up (6 months)
  Distress Thermometer. The distress thermometer is a single-item distress screening scale, which has been shown to be a valid measure of cancer-specific distress among prostate cancer patients and their partners. Participants indicate their current level of distress on an 11-point scale from 0-10 with 0 being no distress and 10 being extreme distress.
Change in quality of life | Baseline and Post Treatment (6 weeks)
  World Health Organization Quality of Life - Brief Form (WHOQOL-BREF). This is a 26-item measure that assesses overall quality of life in four domains of physical health, psychological well-being, social relationships, and environmental well-being. The four domains score with a range from 4-20 with higher scores representing higher quality of life in each domain.
Change in quality of life | Baseline and Follow Up (6 months)
  World Health Organization Quality of Life - Brief Form (WHOQOL-BREF). This is a 26-item measure that assesses overall quality of life in four domains of physical health, psychological well-being, social relationships, and environmental well-being. The four domains score with a range from 4-20 with higher scores representing higher quality of life in each domain.

OTHER OUTCOMES:
Change in Mindfulness | Baseline and Post Treatment (6 weeks)
  Five Facets of Mindfulness questionnaire; Short form, which is a validated, 24-item measure of different aspects of mindfulness. There are five subscales: non-reactivity, observing, acting with awareness, describing, and non-judging. Sub-scale scores range from 5-25 for non-reactivity, acting with awareness, describing, and non-judging, and 5-20 for observing. Higher scores indicate greater levels of the respective facet of mindfulness.
Change in Mindfulness | Baseline and Follow Up (6 months)
  Five Facets of Mindfulness questionnaire; Short form, which is a validated, 24-item measure of different aspects of mindfulness. There are five subscales: non-reactivity, observing, acting with awareness, describing, and non-judging. Sub-scale scores range from 5-25 for non-reactivity, acting with awareness, describing, and non-judging, and 5-20 for observing. Higher scores indicate greater levels of the respective facet of mindfulness.
Mindfulness (moderator) | Baseline
  Five Facets of Mindfulness questionnaire; Short form, which is a validated, 24-item measure of different aspects of mindfulness. There are five subscales: non-reactivity, observing, acting with awareness, describing, and non-judging. Sub-scale scores range from 5-25 for non-reactivity, acting with awareness, describing, and non-judging, and 5-20 for observing. Higher scores indicate greater levels of the respective facet of mindfulness.
Mindfulness (moderator) | Post-Treatment (Week 6)
  Five Facets of Mindfulness questionnaire; Short form, which is a validated, 24-item measure of different aspects of mindfulness. There are five subscales: non-reactivity, observing, acting with awareness, describing, and non-judging. Sub-scale scores range from 5-25 for non-reactivity, acting with awareness, describing, and non-judging, and 5-20 for observing. Higher scores indicate greater levels of the respective facet of mindfulness.
Mindfulness (moderator) | Follow-Up (6 Months)
  Five Facets of Mindfulness questionnaire; Short form, which is a validated, 24-item measure of different aspects of mindfulness. There are five subscales: non-reactivity, observing, acting with awareness, describing, and non-judging. Sub-scale scores range from 5-25 for non-reactivity, acting with awareness, describing, and non-judging, and 5-20 for observing. Higher scores indicate greater levels of the respective facet of mindfulness.
Expectations for treatment (moderator) | Baseline for Treatment Groups
  A 4-item questionnaire, designed for and used in a previous mindfulness-based treatment study for women with provoked vestibulodynia. Scores for each item range from 0-10, with higher scores indicating a greater expectation for the treatment to be effective and greater motivation to complete the treatment and assignments.
Expectations for treatment (moderator) | Post-Treatment (Week 6)
  A 4-item questionnaire, designed for and used in a previous mindfulness-based treatment study for women with provoked vestibulodynia. Scores for each item range from 0-10, with higher scores indicating a greater expectation for the treatment to be effective and greater motivation to complete the treatment and assignments.
Expectations for treatment (moderator) | Follow-Up (6 Months) for Treatment Groups
  A 4-item questionnaire, designed for and used in a previous mindfulness-based treatment study for women with provoked vestibulodynia. Scores for each item range from 0-10, with higher scores indicating a greater expectation for the treatment to be effective and greater motivation to complete the treatment and assignments.
Therapeutic Skills Practice (moderator) | Week 1-4 for Treatment Groups
  This is a questionnaire designed by the experimenters to assess the amount that participants practice the skills taught in treatment daily. Participants will indicate the skills practiced each day, and number of minutes they spent practicing each skill. This will be expressed as total number of minutes or an average of minutes per day.
Therapeutic Skills Practice (moderator) | Follow-Up (6 Months) for Treatment Groups
  This is a questionnaire designed by the experimenters to assess the amount that participants practice the skills taught in treatment. Participants will indicate the skills practiced each day, and number of minutes they spent practicing each skill. This will be expressed as total number of minutes or an average of minutes per day.
Big Five Inventory-10 (moderator) | Baseline
  Big Five Inventory-10. An adapted, brief 10-item measure of personality characteristics. Scores range from 2-10 on the five personality traits of openness to experience, conscientiousness, extroversion, agreeableness, and neuroticism. Higher scores indicate higher levels of the respective trait.
Pre-treatment sexual functioning (moderator) | Baseline
  This is an experimenter derived questionnaire asking participants to indicate if they have a history of sexual dysfunction that preceded their own/their partner's prostate cancer treatments. Items are scored on a range from 0-5, with higher scores denoting greater sexual dysfunction. Total number of items varies as participants are able to specify more dysfunction symptoms.
Time elapsed since treatment (moderator) | Baseline and Follow-Up (6 Months)
  This measure will review date of prostate cancer diagnosis and the time elapsed from treatment to enrollment. This will be reviewed at 6 Months to capture any changes in treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Brotto, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Gordon & Leslie Diamond Health Centre -- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Vancouver Prostate Centre Website — http://www.prostatecentre.com/
- See also: University of British Columbia Sexual Health Lab Website — http://brottolab.med.ubc.ca

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03365518/Prot_SAP_001.pdf